CLINICAL TRIAL: NCT03161717
Title: A Comparative Study of Success Rate, Efficacy, Safety Between Electrical Stimulation-guided Epidural Catheter Placement and the Loss of Resistance Conventional Method for Vaginal Delivery
Brief Title: Efficacy and Safety of Electrical Stimulation-guided Epidural Analgesia for Vaginal Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sang Sik Choi (Other)
Collaborators: Sewoon Medical Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Sang Sik Choi, Professor, Korea University Guro Hospital
Organization: Korea University Guro Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD14043 (RegionalStimⓡ)
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Epidural Analgesia
Keywords: electrical stimulation; vaginal delivery

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural electrical stimulation (EES) (Experimental): n=20
  Interventions: Device: Epidural electrical stimulation (EES)
- Loss of resistance (LOR) (Active Comparator): n=20
  Interventions: Device: Loss of resistance (LOR)

INTERVENTIONS:
Device: Epidural electrical stimulation (EES) — Using loss of resistance technique and electrical stimulation
  Arms: Epidural electrical stimulation (EES)
Device: Loss of resistance (LOR) — Using loss of resistance technique only
  Arms: Loss of resistance (LOR)

SUMMARY:
Forty pregnant women (36 to 41 weeks gestation) will randomly allocate to two groups. Groups will be defined based on the method used to identify the epidural space for epidural anesthesia: the loss of resistance group (n=20) and the epidural electrical stimulation group (n=20). Pain will be assessed using a numerical visual analog scale and maternal satisfaction by a post-partum interview. The success rate of epidural analgesia, maternal satisfaction, and neonatal Apgar scores will be compared between groups.

DETAILED DESCRIPTION:
Investigators will place epidural catheter in the epidural space using loss of resistance technique, and will confirm correct placement of the epidural catheter using electrical stimulation.

Epidural catheter placement, electrical stimulation, and confirmation of response is followed:

Patients will be placed in the left lateral decubitus position. The site will be aseptically prepared and 1% lidocaine will be infiltrated to the skin. An 18-gauge Tuohy needle will be inserted midline of L4/5 interspinous space.

For the Loss of resistance (LOR) group, after identification of the epidural space, the Tuohy needle will be stopped, and a 20-gauge epidural catheter will be advanced through the Tuohy needle.

The same process will be followed for the Epidural electrical stimulation (EES) group. In addition, the epidural space will be confirmed by epidural electrical stimulation using a 20-gauge epidural catheter (RegionalStimTm, Sewoon Medical Co., Ltd, Seoul, Korea, 800 mm) with a conductive guidewire (conductive guidewire, Nitinol, 1100 mm).

After confirming there is no reverse flow of cerebrospinal fluid or blood with aspiration, 3 mL of 1% lidocaine, with 15 mcg of epinephrine (1:200000), will be injected through the epidural catheter as test dose. If there is no response to the test dose, patients will be moved to the delivery room. To control labor pain, a one-time injection containing 50 mcg of fentanyl, 3 mL of 0.75% ropivacaine, and 6 mL of normal saline (total volume 10 mL) will be administered. A continuous infusion of 3 to 10 mL/hour depending on the patient's pain will be used of 75 mcg of fentanyl, 8.5 mL of 0.75% ropivacaine, and 40 mL of normal saline (total volume 50 mL).

Blood pressure (BP), heart rate (HR), oxygen saturation (SpO2), and neurologic assessment findings will be monitored up to 72 hours after labor.

Pain relief in labor is assessed by a change in the visual analogue scale (VAS) score. A 10 point VAS, where 0 is no pain and 10 is unbearable pain, is used to assess pain during labor. The scale is assessed before epidural anesthesia and after epidural anesthesia. Differences in the VAS response we used to assess the efficacy of the epidural anesthesia in decreasing labor pain. Comparison of the change in VAS between groups is used to compare pain control of the two methods. The success of epidural analgesia is defined by sensory block, without motor block, and a decrease in pain score after adequate dosing of epidural medication. Failure of epidural analgesia is defined by a lack of sensory block and a less that 2 point difference on the VAS after adequate dosing of epidural medications.

Patient satisfaction will be evaluated by a postpartum interview. Satisfaction is graded between a score of 1-5, where 1 represent very unsatisfied and 5 represent very satisfied. Patients will indicate a score of 1 to 5.

One- and 5-minute Apgar scores will be compared to assess the effect of epidural electrical stimulation on the neonate. Additional time required for epidural electrical stimulation will be determined by the difference (in seconds) from LOR to identification of the epidural space through electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were at 36 to 41 weeks' gestation and admitted in labor to the university clinic for vaginal delivery were included. Patients were American Society of Anesthesiologists (ASA) physical status of I or II, and were scheduled to receive epidural analgesia

Exclusion Criteria:

* Skin infection at the injection site
* Difficult catheter placement owing to previous lumbar spinal surgery or deformity
* Presence of a hemostatic disorder or use of antiplatelet therapy
* Injection of an analgesic within the previous 12 hours
* Presence of a cardiac pacemaker

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Maternal
Enrollment: 40 (Estimated)
Dates: Start 2015-03-11 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Success rate of epidural analgesia | Up to 6 months
  Evaluation parameter : Accuracy comparison between loss of resistance and epidural electrical stimulation

SECONDARY OUTCOMES:
Maternal satisfaction | Up to 6 months
  Patient satisfaction will be evaluated by a postpartum interview. Satisfaction is graded between a score of 1-5, where 1 represent very unsatisfied and 5 represent very satisfied. Patients will indicate a score of 1 to 5
Neonatal Apgar score | Up to 6 months
  Assessment of neonatal
Procedure-related complications | Up to 6 months
  * Check allergy reaction of anesthetics or chlorohexidine
  * Check whether Insert of local anesthetics to intravascular or not
Minimum electrical current to elicit a response in the epidural electrical stimulation group | Up to 6 months
  * Check stimulation strength that patients begin the feel for the first
  * Check the proper stimulation part of body
Additional time for epidural electrical stimulation | Up to 6 months
  Determined by the difference (in seconds) from loss of resistance(LOR) to identification of the epidural space through electrical stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Sang Sik Choi, MD, PhD, Principal Investigator — Korea University Guro Hiospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva M, Halpern SH. Epidural analgesia for labor: Current techniques. Local Reg Anesth. 2010;3:143-53. doi: 10.2147/LRA.S10237. Epub 2010 Dec 8. PMID 23144567
- [Background] Wantman A, Hancox N, Howell PR. Techniques for identifying the epidural space: a survey of practice amongst anaesthetists in the UK. Anaesthesia. 2006 Apr;61(4):370-5. doi: 10.1111/j.1365-2044.2006.04534.x. PMID 16548958
- [Background] Eappen S, Blinn A, Segal S. Incidence of epidural catheter replacement in parturients: a retrospective chart review. Int J Obstet Anesth. 1998 Oct;7(4):220-5. doi: 10.1016/s0959-289x(98)80042-3. PMID 15321183
- [Background] Hermanides J, Hollmann MW, Stevens MF, Lirk P. Failed epidural: causes and management. Br J Anaesth. 2012 Aug;109(2):144-54. doi: 10.1093/bja/aes214. Epub 2012 Jun 26. PMID 22735301
- [Background] Tsui BC, Tarkkila P, Gupta S, Kearney R. Confirmation of caudal needle placement using nerve stimulation. Anesthesiology. 1999 Aug;91(2):374-8. doi: 10.1097/00000542-199908000-00010. PMID 10443599
- [Background] Tsui BC, Gupta S, Finucane B. Confirmation of epidural catheter placement using nerve stimulation. Can J Anaesth. 1998 Jul;45(7):640-4. doi: 10.1007/BF03012093. PMID 9717595